CLINICAL TRIAL: NCT03244527
Title: Use of BCAA-rich Protein Supplements for Chronic Stroke Patients to Improve the Functional Performance
Brief Title: Use of BCAA-rich Protein Supplements for Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Yen-Nung Lin, Medical doctor of Department of Physical Medicine & Rehabilitation, Taipei Medical University WanFang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N201703029
Record Dates: First submitted 2017-07-21; First posted 2017-08-09 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Stroke
Keywords: BCAA; stroke; mobility
MeSH Terms: conditions — Stroke | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCAA group (Experimental): Participants in the BCAA group take 40g of BCAA supplement before each aerobic exercise session. The interventions include 24 aerobic training sessions. Accordingly, the participants intake 960g of BCAA during a 8-week intervention period.
  Interventions: Dietary Supplement: BCAA supplement; Other: Aerobic exercise
- Control group (Placebo Comparator): Participants in the control group take 40g of placebo before each aerobic training session. The placebo has the same caloric as the BCAA supplement but with different constitution (eg, different percentage of protein, fat and carbohydrate)
  Interventions: Dietary Supplement: BCAA supplement; Other: Aerobic exercise

INTERVENTIONS:
Dietary Supplement: BCAA supplement — Before each exercise session (described later), the research assistant will give subjects 40g of BCAA or placebo supplement according to the treatment assignment and ask them to drink it down right away.
Other: Aerobic exercise — The exercise intervention includes 24 aerobic stationary cycling sessions (30 min/session, 3 session/week, and 8 weeks). The exercise sessions proceed under the supervision and guidance of a therapist.

SUMMARY:
In the past few years, Branched Chain Amino Acid (BCAA) supplements have gradually used on different groups. From training athletes, maintaining functions of healthy elders to preventing disabilities of people that can't do intense exercises. BCAAs are now considered to be able to prevent muscle atrophy and strength loss, also possible to increase strength and muscle mass if combined with resistance exercises. Stroke patients have difficulties with moving, which led to multiple disabilities, are more likely to have sarcopenia and strength loss. Furthermore, reducing the will of moving or walking. Recently, studies showed that combined BCAAs with resistance exercises can effectively increase muscle mass, thus commonly used on training athletes.

Although aerobic exercises are proven to be more likely to improve walking ability of chronic stroke patients than traditional rehabilitation, BCAAs' effects are yet to be proven. Therefore, the aim of this study is to explore if BCAAs combined with moderate intensity exercises can prevent muscle atrophy, loss of strength and cardiopulmonary function.

This is a randomized control trial. Participants are randomly assigned to either experiment or control groups. Both group received aerobic exercise (30 min in a session, 3 days a week, and for 8 weeks). Experiment group received BCAA supplement immediately after the exercise while the control group receive sham product (vitamins). The outcome measurements (including muscle mass, functional measures, and quality of life) are performed before (0-wk) and after (8-wk) the interventions, also after interventions in 3 months and 6 months for follow up.

DETAILED DESCRIPTION:
Setting : inpatient rehabilitation department of Wan-Fang Hospital and Shuang-Ho Hospital Study population : Patients received inpatient treatment or rehabilitation for stroke in Wan-Fang Hospital (WFH) and Shuang-Ho Hospital (SHH).

Study design: controlled trial with randomization Blinding : The patients were blinded by the real or sham bcaa supplements. The assessors who performed the outcome measurements were blinded to the assignment of treatment.

Measurements : DXA(Dual-energy X-ray absorptiometry),CPET(Cardiopulmonary Exercise Testing),6 minute walk test,Timed up and go,Berg balance test,Stroke Specific Quality of Life Scale (SS-QOL).

These measurements (including the clinical and corticomotor excitability assessments) are performed by one researcher who are responsible for the measurements.

Compliance and side effect. The compliance of supplements were investigated. The attendance of treatments (including bcaa supplements and physical therapy sessions) and possible side effect/discomfort were recorded during the interventions by a researcher. He also tries to understand the reason of drop-out from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic stroke>6months
2. Age : 20-75 y
3. Able to walk independently over 30 mins (with or without orthosis)
4. Able to use stationary bike

Exclusion Criteria:

1. Physiological condition not stable, cognitive dysfunction, not able to coordinate with examine or treatments.
2. Not able to exercise due to severe cardiopulmonary dysfunction
3. Malnutrition (MNA<11)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-05 (Actual)

PRIMARY OUTCOMES:
DXA | 8 weeks after intervention
Body fat scale | 8 weeks after intervention

SECONDARY OUTCOMES:
Timed up and go (TUG) | 8 weeks after intervention
Burg Balance Test | 8 weeks after intervention
CPET | 8 weeks after intervention
Stroke Specific Quality of Life Scale(SS-QOL) | 8 weeks after intervention
6 minutes walk test | 8 weeks after intervention

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Shuang-Ho Hospital, New Taipei City
  - WanFang Hospital, Taipei

REFERENCES:
- [Derived] Cheng YH, Wei L, Chan WP, Hsu CY, Huang SW, Wang H, Lin YN. Effects of protein supplementation on aerobic training-induced gains in cardiopulmonary fitness, muscle mass, and functional performance in chronic stroke: A randomized controlled pilot study. Clin Nutr. 2020 Sep;39(9):2743-2750. doi: 10.1016/j.clnu.2019.12.013. Epub 2019 Dec 17. PMID 31879077